CLINICAL TRIAL: NCT05570188
Title: An Investigator-initiated Trial Evaluating the Efficacy and Safety of Anti-CD19 Universal CAR-NK(U-CAR-NK) Cells Therapy Combined With Hematopoietic Stem Cell Transplantation(HSCT) for B Cell Hematologic Malignancies
Brief Title: Anti-CD19 Universal CAR-NK Cells Therapy Combined With HSCT for B Cell Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The PI decides to stop.
Sponsor: Kunming Hope of Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC042
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: B-cell Lymphoma; B-cell Leukemia
Keywords: universal CAR-NK; Hematopoietic Stem Cell Transplantation(HSCT)
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients will get infused with anti-CD19 CAR-NK cells within 1 week after hematopoietic stem cell infusion.
  Interventions: Biological: anti-CD19 UCAR-NK cells

INTERVENTIONS:
Biological: anti-CD19 UCAR-NK cells — Enrolled participants are chosen to receive one of three different dose levels of U-CAR-NK cells:
  Dose level one: 5-10×10^6/kg; Dose level two:1-2×10^7/kg; Dose level three:2-5×10^7/kg.

SUMMARY:
It is a single-center, open-labeled, single-arm, non-randomized investigator-initiated trial evaluating the efficacy and safety of anti-CD19 U-CAR-NK Cells Therapy combined with HSCT for B cell hematologic malignancies.

DETAILED DESCRIPTION:
Who can participate? Patients who were diagnosed with B cell hematologic malignancies and tumor cells expressing CD19.

How to conduct this study? This study is an interventional clinical study. The intervention in the trial is anti-CD19 U-CAR-NK cells, which belong to chimeric antigen receptor modified NK cells. The administration time is 1-7 days after hematopoietic stem cell infusion. Patients were then evaluated for long-term efficacy and safety until 2 years after U-CAR-NK cells infusion.

What are the possible benefits and risks of participating? Benefits: The Dual effect of anti-tumor and anti-infection of NK cells may be used to promote the engraftment of hematopoietic stem cell and better disease control.

Risks: Subjects may have adverse reactions to the treatment. These adverse reactions may include abnormal liver injury, fever, thrombocytopenia, thrombotic microangiopathy, and possibly other unknown adverse reactions.

Where is the study run? Kunming Hope of Health Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with indications for hematopoietic stem cell transplantation;
2. Age ≤75 years old;
3. Confirmed B-cell tumor and tumor cells expressing CD19；
4. Expected survival time >12 weeks;
5. ECOG score is 0-2;
6. Adequate liver , kidney and cardiopulmonary function;
7. Willingness to complete the informed consent process and to comply with study procedures and visit schedule.

Exclusion Criteria:

1. Had received NK cell therapy or other genetically modified cell therapy within 1 year before screening;
2. At least 14 days or at least 5 half-lives of antitumor therapy had elapsed before screening;
3. Patients who had undergone hematopoietic stem cell transplantation (ASCT), allogeneic hematopoietic stem cell transplantation (HSCT), or solid organ transplantation within 12 weeks before screening; Grade 2 or higher GVHD requiring immunosuppressive therapy occurred within 2 weeks before screening;
4. Patients with atrial or ventricular lymphoma or need urgent treatment due to tumor mass such as intestinal obstruction or vascular compression;
5. Have received live attenuated vaccine within 6 weeks before rinsing;
6. Had a cerebrovascular accident or seizure within 6 months before screening;
7. History of deep venous thrombosis or pulmonary embolism within 6 months before screening;
8. A history of myocardial infarction, bypass or stent bypass, unstable angina, or other clinically significant heart disease within 12 months prior to screening;
9. Previous history of Alzheimer's disease;
10. Autoimmune diseases leading to end-organ damage or requiring systemic immunosuppression (e.g. Crohns, rheumatoid arthritis, systemic lupus erythematosus) within 2 years prior to screening;
11. There are uncontrollable infections;
12. Women who are pregnant or breastfeeding; Or women of childbearing age who have positive pregnancy tests during the screening period; Male or female patients who did not wish to use contraception from the time of signing the informed consent to 1 year after receiving the NK cell infusion;
13. Conditions that other researchers deemed inappropriate for participating in the study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included. Description, time, classification, and outcome of AE events resulted from the investigational medical product, delivery method, or emergency measures will be recorded in the case report form.

SECONDARY OUTCOMES:
Granulocyte implantation time | Up to 1 month after infusion
  Time from hematopoietic stem cell transfusion to peripheral blood granulocyte count >0.5×10^9/L for 3 consecutive days.
Platelet implantation time | Up to 1 month after infusion
  Time from hematopoietic stem cell transfusion to peripheral blood platelet count >20×10^9/L for 7 consecutive days.
Red blood cell implantation time | Up to 1 month after infusion
  Time from hematopoietic stem cell transfusion to peripheral blood hemoglobin count >70g/L.
Duration of remission (DOR) | Up to 24 weeks after infusion
  Duration of remission (DOR) refers to the time from the first assessment of CR or PR of the tumor to the first assessment of disease recurrence or progression or death from any cause.
Disease control rate (DCR) | Up to 24 weeks after infusion
  Disease control rate (DCR) are defined as the percentage of patients who have achieved complete response, partial response or stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Overall survival (OS) | Up to 24 weeks after infusion
  Overall survival (OS) refers to the time from the time the patient received an infusion of CAR-NK cells until death (from any cause).
Progression-free survival (PFS) | Up to 24 weeks after infusion
  Progression-free survival (PFS) refers to the time from the start of treatment with CAR-NK cells to the first progression of disease or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, Principal Investigator — Kunming Hope of Health Hospital
Locations (1):
- Kunming Hope of Health Hospital, Kunming, Yunnan, China